CLINICAL TRIAL: NCT06938269
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single-and Multiple-Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of MWN109 Tablets in Healthy Adult Participants
Brief Title: A Study to Evaluate MWN109 Tablets in Healthy Adult Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Minwei Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MWN109-T-101
Record Dates: First submitted 2025-04-14; First posted 2025-04-22 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Overweight or Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Participants in SAD cohorts will be randomized to receive a single dose of MWN109 tablet or placebo across 4 cohorts. Participants in MAD cohorts will be randomized to receive MWN109 tablet or placebo once daily for 28 days in cohorts B1 and B2, 30 days in cohort B3.
  Interventions: Drug: Placebo
- MWN109 tablets (Active Comparator): Participants in SAD cohorts will be randomized to receive a single dose of MWN109 tablet or placebo across 4 cohorts. Planned dosage per cohorts are A1:7.5mg, A2:15mg, A3:30mg, A4:45mg.
  Participants in MAD cohorts will be randomized to receive MWN109 tablet or placebo once daily for a total of 28 days in cohorts B1 and B2, 30 days in cohort B3. Initiation and dose levels of MAD cohorts will be determined in the safety review and dose escalation meeting by the Safety Review Committee based on the review of safety, tolerability, and PK data from SAD part. The target doses could be 15mg, 30mg and 45 mg.
  Interventions: Drug: MWN109 tablet

INTERVENTIONS:
Drug: MWN109 tablet — Strength: 4mg, 7.5mg, 15mg, 30mg, and 45 mg; Administration: Oral.
  Arms: MWN109 tablets
Drug: Placebo — Administration: Oral.
  Arms: Placebo

SUMMARY:
This is a Phase 1, randomized, double-blind, placebo-controlled, single-and-multiple ascending dose study in which the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and immunogenicity of orally administered MWN109 tablets will be assessed in healthy adult participants.

DETAILED DESCRIPTION:
Approximately 60 healthy volunteers are expected to be enrolled into this study. The study will consist of 2 parts: a single ascending dose (SAD) part and a multiple ascending dose (MAD) part.The SAD part will be a single-dose, sequential-cohort study. The MAD Part will be a multiple-dose, sequential-cohort study. Initiation and dose levels of MAD Part will be determined in the safety review and dose escalation meeting by the Safety Review Committee based on the review of safety, tolerability, and PK data from SAD Part.

The entire study duration per participant is estimated to be a maximum of 8 weeks for the single ascending dose (SAD) part and 12 weeks for the multiple ascending dose (MAD) part. The end of study is defined as the date of the last visit of the last participant in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged 18 to 60 years (inclusive) at the time of signing the informed consent (Caucasians should be no less than 80% since the implementation of Protocol Clarification Letter #2, dated 02 Sep 2025).
2. [Part A: SAD] Body mass index (BMI) of 19.0 to 40.0 kg/m2 (inclusive) with body weight > 65.0 kg and <130.0 kg. [Part B: MAD] BMI of 27.0 to 45.0 kg/m2 (inclusive) with body weight > 65.0 kg and <130.0 kg.
3. Stable body weight within 3 months before screening (defined as self-reported change < 5%).
4. Resting heart rate (supine) ≥ 45 bpm and ≤ 90 bpm with a single 12-lead ECG at Screening. If the heart rate is > 90 or < 45 bpm, it is to be repeated 2 more times (separated by at least 2 min) and the average of the 3 heart rate values is to be used to determine the participant's eligibility.
5. Females of childbearing potential and males who are not surgically sterile (>180 days since vasectomy with no viable sperm) will agree to use contraception from Screening until 4 months after the last administration, OR females of non-reproductive potential as defined below:

   * Postmenopausal as defined as:

     * No menses for at least 12 months; OR
     * No menses for at least 12 months AND with a follicle-stimulating hormone level > 40 IU/L or according to the definition of "postmenopausal range" for the laboratory involved; OR
   * History of hysterectomy; OR
   * History of bilateral oophorectomy
6. Male participants must agree to refrain from sperm donation and females should refrain from ova donation from Screening until 4 months after the last administration.
7. Willing to maintain current general diet and physical activity regimen, except for the physical activity in the 72 h before each blood sample collection for the clinical laboratory analysis, which should not be strenuous, and willing to be restrained from alcohol and smoking during the study period.
8. Able to comprehend and willing to sign an informed consent form (ICF) and to abide by all study requirements and restrictions.

Exclusion Criteria:

1. Significant history or clinical manifestation of any cardiovascular, metabolic, allergic, endocrine, renal, hepatic, gastrointestinal, hematological, pulmonary, respiratory, dermatological, neurological, gynecological, psychiatric disorders, as determined by the Principal Investigator (or delegate).
2. Screening blood pressure in supine outside the ranges 90-159 mmHg systolic, 50-95 mmHg diastolic. If abnormal blood pressure is observed, the blood pressure is to be repeated 2 more times, and the average of the 3 blood pressure values is to be used to determine the participant eligibility.
3. History of insulinoma, or has an event of blood glucose < 2.8 mmol/L within 1 year prior to Screening, or with ≥ 3 times of hypoglycemia symptoms within 3 months prior to Screening.
4. History of febrile illness within 7 days prior to the first dose of IP or participants with evidence of active infection.
5. Any of the following:

   1. QTcF > 450 msec confirmed by repeat measurement;
   2. QRS duration > 120 msec confirmed by repeat measurement;
   3. PR interval > 220 msec confirmed by repeat measurement. Notes: Regarding a), b) and c), ECG is to be repeated 2 more times when out-of-range and the average of the values is to be used to determine the participant eligibility;
   4. Findings which would make QTc measurements difficult or QTc data uninterpretable;
   5. History of additional risk factors for torsades de pointes (e.g., heart failure, hypokalemia, family history of long QT syndrome).
6. Known history or family history of thyroid C-cell tumor/carcinoma, multiple endocrine neoplasia syndrome type 2 (MEN2), thyroid dysfunction or thyroid hormone abnormality.
7. History of diabetes mellitus or clinical evidence of diabetes (e.g., hemoglobin A1c ≥ 6.5%, fasting plasma glucose ≥ 126 mg/dL [7.0 mmol/L]) at Screening, non-fasting plasma glucose ≥ 200 mg/dL (11.1 mmol/L) at Screening, or use of any hypoglycemic drugs during Screening or within 3 months prior to Screening.
8. History of acute or chronic pancreatitis, symptomatic gallbladder disease, pancreatic injury and other high-risk factors that may lead to pancreatitis.
9. With any of following laboratory abnormality at screening and confirmed by a single repeat at the discretion of the Principal Investigator (or delegate):

   a) Elevation in serum amylase or lipase (> 1.5 × upper limit of normal [ULN]). b) Have serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 1.5 × ULN or total bilirubin >1.5 × ULN.

   c) Have serum triglycerides (TG) ≥ 5.65 mmol/L (500 mg/dL) at Screening. d) Estimated glomerular filtration rate (eGFR) < 80 mL/min/1.73m2 by Cockcroft-Gault equation as below: (140 - age) × mass (kg)/72 × creatinine (mg/dL); multiply by 0.85 if female.
10. Untreated or uncontrolled hypothyroidism/hyperthyroidism defined as thyroid-stimulating hormone > 6 mIU/L or < 0.4 mIU/L.
11. History of clinically significant (in the opinion of the Principal Investigator or delegate) abnormal gastric emptying (e.g., gastric outlet obstruction, gastroparesis), chronic gastrointestinal diseases (e.g., having active ulcer within 6 months prior to Screening, active gastritis or esophagitis, or gastroesophageal reflux disease, irritable bowel disease or severe inflammatory bowel disease).
12. Presence of clinically significant acute gastrointestinal symptoms (e.g., nausea, vomiting, heartburn or diarrhoea) or malabsorptive states (celiac disease, lactose intolerance or chronic pancreatitis), as judged by the Principal Investigator (or delegate).
13. Any history or plan of gastrointestinal surgery excluding appendectomy.
14. Positive hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV-Ab), or human immunodeficiency virus (HIV-1 and HIV-2) antibodies.
15. Any history of severe psychiatric disorder such as major depressive disorder, bipolar disorder, and schizophrenia, or history of suicidal ideation, behavior or attempts or other psychiatric disorder.
16. History of alcoholism or drug/chemical abuse within 1 year prior to D-1.
17. Alcohol consumption of > 21 units per week for males and > 14 units per week for females, on average. One unit of alcohol equals 1/2 pint (285 mL) of beer, 1 glass (125 mL) of wine, or 1/6 gill (25 mL) of spirits.
18. Positive alcohol breath test result or positive urine drug screen (confirmed by repeat) during the Screening period.
19. Daily use of more than 10 cigarettes/day (on average), or 2 cigars/day (on average), or equivalent use of any nicotine-containing product within 6 weeks prior to Screening.
20. Participant is unwilling to refrain from strenuous exercise (e.g., heavy lifting, weight training, and aerobics) for 72 h prior to each blood collection for clinical laboratory tests.
21. Females of pregnant or lactating, or those with a positive pregnancy test at Screening.
22. Intolerance to venipuncture for blood sampling or history of fainting at blood drawing or sight of blood, unless deemed acceptable by the Principal Investigator (or delegate).
23. Long-term use of drugs directly affecting the gastrointestinal motility (including but not limited to mosapride, cisapride) or gastrointestinal surgery within 12 weeks prior to Screening and are inappropriate for participation in this clinical study as assessed by the Principal Investigator (or delegate).
24. History of severe Types I-IV hypersensitivity reactions, anaphylaxis, cytokine release syndrome, atopic individuals, or allergic reactions to multiple drugs. If the Principal Investigator (or delegate) is considering enrolling a participant with multiple drug allergies, agreement with the Medical Monitor should be sought.
25. History of or suspected allergy or hypersensitivity to the IP or its components.
26. Use or intend to use any prescription medications/products other than hormone replacement therapy, oral, implantable, transdermal, injectable, or intrauterine contraceptives within 14 days prior to dosing, unless deemed acceptable by the Principal Investigator (or delegate)and agreement with the Sponsor.
27. Use or intend to use slow-release medications/products considered to still be active within 14 days prior to D-1, unless deemed acceptable by the Principal Investigator (or delegate).
28. Use of any nonprescription medications/products including vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations within 7 days prior to D-1 or during the study, unless deemed acceptable by the Principal Investigator (or delegate) and agreement with Sponsor, with the exception of paracetamol/acetaminophen (maximum 2 g per day for up to 3 days) and topically applied medications which is permitted up to 48 h prior to dosing.
29. Participants with a history of infectious diseases (which may affect the ability of the participant to participate in the study at the discretion of the Principal Investigator or delegate), severe trauma, or major surgical operation within 4 weeks prior to Screening.
30. Have been vaccinated within 4 weeks prior to Screening or plan to have vaccination during the study.
31. Donation of blood or massive blood loss (> 450 mL) OR receipt of blood products within 12 weeks prior to Screening, plasma from 2 weeks prior to Screening, and platelets from 6 weeks prior to Screening.
32. Participation in a clinical study involving administration of an investigational agent/device or vaccine (new chemical entity) within 30 days or 5 half-lives, or having received a biological product within 12 weeks prior to Screening.
33. Poor peripheral venous access.
34. Are investigative site personnel directly affiliated with this study and their immediate families. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.
35. The presence of clinically significant physical examination, vital sign, drug, or ECG findings at Screening or baseline or laboratory findings at Screening that, in the opinion of the Principal Investigator (or delegate) or Medical Monitor, may interfere with any aspect of study conduct or interpretation of results.
36. Are deemed unsuitable by the Principal Investigator (or delegate) for any other reason.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Incidence of treatment emergent adverse events (TEAEs) following treatment administration | SAD: Up to Day 22; MAD: Up to Day 56 (Cohorts B1 and B2) or Day 58 (Cohort B3) post first dose administration
Number of participants with change in laboratory parameters following treatment administration | SAD: Up to Day 22; MAD: Up to Day 56 (Cohorts B1 and B2) or Day 58 (Cohort B3) post first dose administration
  Clinical safety laboratory measures include urine drug screening, alcohol breath test, serum virology, pregnancy test, chemistry, hematology, urinalysis and thyroid function.
Number of participants with change in 12-lead ECG following treatment administration | SAD: Up to Day 22; MAD: Up to Day 56 (Cohorts B1 and B2) or Day 58 (Cohort B3) post first dose administration
Number of participants with change in Vital signs following treatment administration | SAD: Up to Day 22; MAD: Up to Day 56 (Cohorts B1 and B2) or Day 58 (Cohort B3) post first dose administration
  Vital signs including pulse rate, respiratory rate, supine blood pressure and tympanic body temperature.
Incidence of anti-drug antibody (ADA) formation following treatment administration | SAD: Up to Day 22; MAD: Up to Day 56 (Cohorts B1 and B2) or Day 58 (Cohort B3) post first dose administration
Number of participants with change in physical examinations following treatment administration | SAD: Up to Day 22; MAD: Up to Day 56 (Cohorts B1 and B2) or Day 58 (Cohort B3) post first dose administration

SECONDARY OUTCOMES:
PK parameters- Cmax: maximum observed concentration | SAD: Up to Day 22; MAD: Up to Day 56 (Cohorts B1 and B2) or Day 58 (Cohort B3) post first dose administration
PK parameters- Tmax: time to reach maximum concentration | SAD: Up to Day 22; MAD: Up to Day 56 (Cohorts B1 and B2) or Day 58 (Cohort B3) post first dose administration
PK parameters- t1/2: half-life | SAD: Up to Day 22; MAD: Up to Day 56 (Cohorts B1 and B2) or Day 58 (Cohort B3) post first dose administration
PK parameters- AUC0-inf: area under the concentration-time curve from time zero to the theoretical infinite time | SAD: Up to Day 22; MAD: Up to Day 56 (Cohorts B1 and B2) or Day 58 (Cohort B3) post first dose administration
PK parameters- AUC0-t: area under the concentration-time curve from time zero to the time of the last quantifiable concentration | SAD: Up to Day 22; MAD: Up to Day 56 (Cohorts B1 and B2) or Day 58 (Cohort B3) post first dose administration
PK parameters- AUC0-168h: area under the concentration-time curve from time zero to 168 h post dose | SAD: Up to Day 22; MAD: Up to Day 56 (Cohorts B1 and B2) or Day 58 (Cohort B3) post first dose administration
PK parameters- CL/F: apparent clearance | SAD: Up to Day 22; MAD: Up to Day 56 (Cohorts B1 and B2) or Day 58 (Cohort B3) post first dose administration
PK parameters- Vd/F: apparent volume of distribution | SAD: Up to Day 22; MAD: Up to Day 56 (Cohorts B1 and B2) or Day 58 (Cohort B3) post first dose administration
PK parameters- MRT: mean residence time | SAD: Up to Day 22; MAD: Up to Day 56 (Cohorts B1 and B2) or Day 58 (Cohort B3) post first dose administration
PK parameters- terminal elimination rate constant | SAD: Up to Day 22; MAD: Up to Day 56 (Cohorts B1 and B2) or Day 58 (Cohort B3) post first dose administration

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - CMAX Clinical Research, Adelaide, South Australia
  - Veritus Research, Bayswater, Victoria

IPD SHARING:
Plan to Share IPD: No